CLINICAL TRIAL: NCT06305975
Title: Blunt Fascial vs. Veress Needle Peritoneal Entry in Laparoscopic Gynecologic Surgery: A Randomized Controlled Trial
Brief Title: Blunt Fascial vs. Veress Needle Peritoneal Entry in Laparoscopic Gynecologic Surgery
Acronym: BluntFascial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Raanan Meyer, Principal Investigator, Cedars-Sinai Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00003169
Record Dates: First submitted 2024-02-22; First posted 2024-03-12 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Laparoscopic Surgery
Keywords: Abdominal entry; Laparoscopy; Insufflation time; Postoperative pain; Safety
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blunt fascial entry (Experimental): The blunt fascial entry technique will be used for patients in this arm
  Interventions: Procedure: Blunt fascial abdominal entry
- Veress needle entry technique (Active Comparator): The Veress needle entry technique will be used for patients in this arm
  Interventions: Procedure: Veress needle abdominal entry

INTERVENTIONS:
Procedure: Blunt fascial abdominal entry — Blunt fascial entry technique description: a 5 mm incision is made in the umbilicus. Next, a curved Kelly forceps is used to open the fascia, and, if possible, the peritoneum. The Kelly forceps are then used to expand the opening to a 10 mm diameter. A 5 mm trocar is placed into the fascial hole and used to quickly insufflate the abdomen to 15 mm Hg. Once the abdomen is fully insufflated, a 10 mm trocar is placed using optical guidance.
  Arms: Blunt fascial entry
Procedure: Veress needle abdominal entry — Veress needle abdominal entry technique description: a 5 mm incision is made in the umbilicus. Next, a Veress needle is used to enter the peritoneal cavity and inflate the abdomen to 15 mm Hg. Once the abdomen is fully insufflated, a 10 mm trocar is placed using optical guidance.
  Arms: Veress needle entry technique

SUMMARY:
This study aims to investigate the effect of two peritoneal entry techniques on intraoperative and post-operative outcomes among patients undergoing laparoscopic surgery with a minimally invasive gynecologic surgeon. Patients will be randomized to either blunt fascial or veress needle peritoneal entry. Insufflation times, failed entries, complications and post-operative pain scores will be collected.

The investigators hypothesize that the blunt entry technique will be associated with shorter insufflation times and similar intraoperative and postoperative outcomes compared with the veress needle entry technique.

Primary Objective: To evaluate the insufflation times and success upon peritoneal entry according to peritoneal entry technique.

Secondary Objectives: To evaluate the surgical outcomes and patients pain scores according to peritoneal entry technique.

DETAILED DESCRIPTION:
This will be a single-center, single-blinded randomized controlled trial evaluating the impact of peritoneal entry technique on insufflation times, entry failure, post-operative pain and surgical outcomes among patients undergoing laparoscopic gynecologic surgery. The investigators hypothesize that the blunt fascial entry technique will be associated with shorter insufflation times with no effect on other surgical outcomes. The study will include 2 groups corresponding to the entry techniques: blunt facial entry and Veress needle entry. Participants will be 1:1 allocated to each technique by block randomization.

Blunt fascial entry technique description: a 5 mm incision is made in the umbilicus. Next, a curved Kelly forceps is used to open the fascia, and, if possible, the peritoneum. The Kelly forceps are then used to expand the opening to a 10 mm diameter. A 5 mm trocar is placed into the fascial hole and used to quickly insufflate the abdomen to 15 mm Hg. Once the abdomen is fully insufflated, a 10 mm trocar is placed using optical guidance.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. 18 years of age or older
4. Undergoing conventional laparoscopic surgery at Cedars-Sinai Medical Center with a surgeon in the Minimally Invasive Gynecologic Surgery division.

Exclusion Criteria:

1. Pregnancy
2. Urgent/non-scheduled surgery
3. Non-eligible for umbilical entry

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03-22 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Insufflation time | Intraoperative
  The time it takes to insufflate the abdominal cavity to 15 mm Hg.
Success upon peritoneal entry | Intraoperative
  Successful abdominal entry in the first trial

SECONDARY OUTCOMES:
Intraoperative complications | Intraoperative
  - Intraoperative complications upon peritoneal entry
Postoperative complications | Postoperative period within 30 days of surgery
  Any postoperative complications
Patients pain scores | Day of surgery, postoperatively and before discharge
  * First reported pain score in PACU using the numerical rating scale (0-10).
  * Last reported pain score in PACU prior to discharge using the numerical rating scale (0-10).
Analgesics use | Day of surgery, postoperatively and before discharge
  - Total analgesic requirements in PACU
Length of hospital stay | Day of surgery, postoperatively and before discharge. In rare cases, hospital stay will be longer than one day.
  - Length of stay- from arrival to PACU to discharge home)

CONTACTS AND LOCATIONS:
Overall Officials: Raanan Meyer, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ahmad G, Baker J, Finnerty J, Phillips K, Watson A. Laparoscopic entry techniques. Cochrane Database Syst Rev. 2019 Jan 18;1(1):CD006583. doi: 10.1002/14651858.CD006583.pub5. PMID 30657163
- [Background] Jansen FW, Kapiteyn K, Trimbos-Kemper T, Hermans J, Trimbos JB. Complications of laparoscopy: a prospective multicentre observational study. Br J Obstet Gynaecol. 1997 May;104(5):595-600. doi: 10.1111/j.1471-0528.1997.tb11539.x. PMID 9166204
- [Background] Makai G, Isaacson K. Complications of gynecologic laparoscopy. Clin Obstet Gynecol. 2009 Sep;52(3):401-11. doi: 10.1097/GRF.0b013e3181b0c080. PMID 19661756
- [Background] Molloy D, Kaloo PD, Cooper M, Nguyen TV. Laparoscopic entry: a literature review and analysis of techniques and complications of primary port entry. Aust N Z J Obstet Gynaecol. 2002 Aug;42(3):246-54. doi: 10.1111/j.0004-8666.2002.00246.x. PMID 12230057
- [Background] Azevedo JL, Azevedo OC, Miyahira SA, Miguel GP, Becker OM Jr, Hypolito OH, Machado AC, Cardia W, Yamaguchi GA, Godinho L, Freire D, Almeida CE, Moreira CH, Freire DF. Injuries caused by Veress needle insertion for creation of pneumoperitoneum: a systematic literature review. Surg Endosc. 2009 Jul;23(7):1428-32. doi: 10.1007/s00464-009-0383-9. Epub 2009 Mar 5. PMID 19263124
- [Background] Jiang X, Anderson C, Schnatz PF. The safety of direct trocar versus Veress needle for laparoscopic entry: a meta-analysis of randomized clinical trials. J Laparoendosc Adv Surg Tech A. 2012 May;22(4):362-70. doi: 10.1089/lap.2011.0432. Epub 2012 Mar 16. PMID 22423957
- [Background] Krishnakumar S, Tambe P. Entry complications in laparoscopic surgery. J Gynecol Endosc Surg. 2009 Jan;1(1):4-11. doi: 10.4103/0974-1216.51902. PMID 22442503
- [Background] Kendrick DB, Strout TD. The minimum clinically significant difference in patient-assigned numeric scores for pain. Am J Emerg Med. 2005 Nov;23(7):828-32. doi: 10.1016/j.ajem.2005.07.009. PMID 16291435
- [Background] Cepeda MS, Africano JM, Polo R, Alcala R, Carr DB. What decline in pain intensity is meaningful to patients with acute pain? Pain. 2003 Sep;105(1-2):151-7. doi: 10.1016/s0304-3959(03)00176-3. PMID 14499431
- [Background] Foley CE, Ryan E, Huang JQ. Less is more: clinical impact of decreasing pneumoperitoneum pressures during robotic surgery. J Robot Surg. 2021 Apr;15(2):299-307. doi: 10.1007/s11701-020-01104-4. Epub 2020 Jun 22. PMID 32572753